CLINICAL TRIAL: NCT06607042
Title: BEDIT-RCT: Randomized Controlled Study on the Effectiveness of Berlin Dissexuality Therapy as Part of the Model Project in Accordance With §65d German Social Security Code V
Brief Title: Study on the Effectiveness of Berlin Dissexuality Therapy as Part of the Model Project in Accordance With §65d SBG V
Acronym: BEDIT-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Hannover Medical School (Other); Heinrich-Heine University, Duesseldorf (Other); Klinikum Bamberg (Other); Universitätsklinikum Kiel (Unknown); University Medical Center Mainz (Other); Uniklinikum Giessen und Marburg (Unknown); University Hospital Ulm (Other); Universitätsklinikum Leipzig (Other); University Hospital Regensburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Klaus Michael Beier, Director, Institute for Sexual Research and Sexual Medicine, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402913; 402913 (Other: ChariteU)
Record Dates: First submitted 2024-09-13; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Paedophilia; Hebephilia
Keywords: Paedophilia; Hebephilia; Child Abuse Images; Sexual Offending
MeSH Terms: conditions — Pedophilia | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group receives treatment
  Interventions: Behavioral: Psychotherapy
- Waitlist Control-group (No Intervention): This group consists of individuals randomized to the waitlist condition

INTERVENTIONS:
Behavioral: Psychotherapy — Psychotherapy according to the Berlin Dissexuality Therapy (BEDIT)
  Arms: Intervention Group

SUMMARY:
The main goal of this clinical trial is to learn if psychotherapy works to reduce consumption of child abuse imagages.

ELIGIBILITY:
Inclusion Criteria:

* Age at first presentation minimum 18 years
* Voluntary consent to participation on the part of the participant
* At the time of inclusion, no contact with the justice system (ongoing investigation, ongoing criminal proceedings, ongoing prison sentence) due to sexually abusive behavior towards children
* Sexually conspicuous behavior and/or fantasies or impulses that indicate the presence of a pedophilic and/or hebephilic preference disorder.
* An offer of treatment is made when a suspected diagnosis is confirmed or the diagnosis is confirmed
* Feared or recent use of abusive images
* Sufficient knowledge of German
* Voluntary participation in the study and checking the checkbox in the informed consent form before starting participation

Exclusion Criteria:

* Age under 18 years
* Lack of consent on the part of the patient
* Exclusion of the presence of a pedophilic and/or hebephilic preference disorder
* Current legal status in the sense of an ongoing investigation or criminal proceedings due to sexually assaultive behavior towards children
* Severe comorbidities: unstable psychotic disorder, organic brain damage, reduced intellectual capacity (IQ below 70), untreated drug or alcohol addiction or persistent harmful use
* Current risk of child sexual abuse and or child sexual abuse that occurred less than 15 years before the start of the study
* An antiandrogenic medication or an opiate antagonist, during therapy start taking a serotonin reuptake inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Abstinence | From enrollment to the end of treatment 12 - 18 weeks
  Abstinence rates for the consumption of abusive images

SECONDARY OUTCOMES:
Frequency of abstinence rates | From enrollment to the end of treatment 12 - 18 weeks
  Frequency of abstinence rates for the use of child abuse images
Sexual preoccupation | From enrollment to the end of treatment 12 - 18 weeks
  Hypersexual Behavior Inventory - 19, Total Sexual Outcomes
  * 19 Items, rated on a scale from 1 (never) bis 5 (very often)
  * No reverse-coded items
  * Unweighted summation
  * minimum = 19, maximum = 95
  * Higher scores indicate more frequent or intense hypersexual behavior (negative outcome)
Cognitive distortions about child sexual abuse | From enrollment to the end of treatment 12 - 18 weeks
  Attitudes conducive to child sexual abuse measured by Bumby Molest Scale
  * 38 items, rated on a scale from 1 (strongly disagree) to 4 (strongly agree)
  * No reverse-coded items
  * Unweighted summation
  * minimum = 38, maximum = 152
  * Higher scores indicate a greater extent of cognitive distortions (negative outcome)
Emotion regulation | From enrollment to the end of treatment 12 - 18 weeks
  Emotion regulation measured by Coping Inventory for Stressful Situations - Short Form
  * 24 items, rated on a scale from 1 (not at all typical) to 5 (very typical)
  * No reverse-coded items
  * Unweighted summation
  * 3 subscales (task-oriented, emotion-oriented, avoidance): minimum = 8, maximum = 40 for each
Mental Health | From enrollment to the end of treatment 12 - 18 weeks
  Mental health measured by Hospital Anxiety and Depression Scale
  * Two subscales (Anxiety and Depression), each with 7 items, rated from 0 (no symptoms) to 3 (severe symptoms)
  * Unweighted summation
  * minimum = 0, maximum = 21 per subscale; cutoff score = 11
  * Even-numbered items pertain to the Depression subscale, odd-numbered items to the Anxiety subscale
  * Items 1, 3, 5, 6, 8, 10, 11, 13 are reverse-coded
General well-being | From enrollment to the end of treatment 12 - 18 weeks
  General well-being measured by European Health Interview Survey - Quality of Life
  * 8 items, rated on a scale from 1 (not at all) to 5 (completely)
  * No reverse-coded items
  * Unweighted summation
  * minimum = 8, maximum = 40
  * Higher scores represent better quality of life

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid, R. C., Garos, S. & Carpenter, B. N. (2011). Reliability, Validity, and Psychometric Development of the Hypersexual Behavior Inventory in an Outpatient Sample of Men. Sexual Health & Compulsivity, 18(1), 30-51. https://doi.org/10.1080/10720162.2011.555709
- [Background] Bumby, K. M. (1996). Assessing the Cognitive Distortions of Child Molesters and Rapists: Development and Validation of the MOLEST and RAPE Scales. Sexual Abuse, 8(1), 37-54. https://doi.org/10.1177/107906329600800105
- [Background] Endler, N. S., & Parker, J. D. A. (1999). Coping Inventory for Stressful Situations--Short Form (CISS-SF) [Database record]. APA PsycTests.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Schmidt S, Muhlan H, Power M. The EUROHIS-QOL 8-item index: psychometric results of a cross-cultural field study. Eur J Public Health. 2006 Aug;16(4):420-8. doi: 10.1093/eurpub/cki155. Epub 2005 Sep 1. PMID 16141303